CLINICAL TRIAL: NCT05441735
Title: The Effectiveness of Digital Care-plan for Improving Long-term Care 2.0 Service Activation Proportion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CHANG HUI PING, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHANG HUI PING
Record Dates: First submitted 2022-06-07; First posted 2022-07-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Digital Care-plan; Long-term Care; Activation Proportion; Case Management, APP(Application)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): will have access to information on the Long-Term Care Plan 2.0 through the app-based digital care program, while the
  Interventions: Combination Product: APP
- control group (No Intervention): will only have access to information on the Long-Term Care Plan 2.0 through conventional paper-based media.

INTERVENTIONS:
Combination Product: APP — APP as an instructional tool for visiting health education
  Arms: experimental group

SUMMARY:
Digital tools can potentially improve the public's reception to and understanding of long-term care information, which will be significantly helpful for long-term care workers and effectively increase the coverage provided by long-term care services. The results of this study could be used to further explore the feasibility of service digitization in the field of long-term care, as well as the integration of technology and professional knowledge to facilitate access to long-term care resources in a modern setting.

DETAILED DESCRIPTION:
Background The number of care recipients served by the 10-Year Long-Term Care Plan 2.0 has grown by approximately 44% since its implementation in 2017. However, only about 228,000 individuals were evaluated by care centers from January to November 2018. This indicates that long-term care services had achieved a service coverage of 29.8% for January-November 2018, serving less than 30% of the individuals who need long-term care. Research on the reasons for not using such services has revealed that the public has limited access to and understanding of information relating to long-term care resources, making it difficult for people draw the connection between their needs and long-term care services.

Aim The study will involve the development of an app-based digital care program, in the hope of enhancing the public's access to and understanding of long-term care information and expanding the coverage realized by long-term care.

Method The study is a two-group randomized controlled trial with an expected sample of 76 participants, and the app-based digital care program will serve as the intervention tool in this study. The experimental group will have access to information on the Long-Term Care Plan 2.0 through the app-based digital care program, while the control group will only have access to information on the Long-Term Care Plan 2.0 through conventional paper-based media. Data collection is then conducted using a pre- and post-test approach and through the administration of a structured questionnaire. The data collected include the participants' willingness to use long-term care services, their attitudes toward long-term care services, and their service use behavior. For the experimental group, an additional survey was also conducted to assess their satisfaction with the use the app-based digital care program to access information, with the aim of examining the effectiveness of the program when used by new Long-Term Care Plan 2.0 cases.

ELIGIBILITY:
Inclusion Criteria:

* Those who meet the eligibility requirements for long-term care services:
* Those who are over 65 years old.
* Those who have no primary caregiver and who have clear consciousness and cognition, who can converse in Mandarin and Taiwanese, who can fill in the questionnaire, or who can
* The researcher read out word for word, filled in after oral answer, and agreed to participate in this researcher.

Primary Caregiver:

* Those who mainly assist the disabled in activities of daily living and provide the most common daily activities for the family
* The caregivers in terms of motor function, or those who are identified as the main caregivers by the disabled, can fill in the questionnaire, or the researchers can read them out verbatim, and fill in the answers after their oral answers.

Exclusion Criteria:

* Those who are not eligible for long-term care services.
* Those who have used the long-term photo 2.0 service.
* Those who cannot operate 3C products or surf the Internet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
using a pre- and post-test approach and through the administration of a structured questionnaire. | 2 months
  This research tool looks forward to understanding long-term care service users, their willingness to use long-term care 2.0 services,
  There are 18 questions in total, including the following topics:
  1. Basic attribute information.
  2. Willingness to activate the service: The higher the score, the higher the willingness to enable the service, with a total score of 25 points.
  3. Attitudes in service use: The higher the score, the closer to a reasonable and appropriate attitude, the higher the score (5 points), and the lower the score (1 point), the total score is 35 points.
  4. Service usage behavior: The answer is based on a five-point Likert Scale (1-5 points). The higher the score, the higher the understandiThe total score is 55 points.

SECONDARY OUTCOMES:
Satisfaction with the use of the app digital care plan (visual analog scale) | 2 months
  Mainly for the experimental group after using the App digital care program for 8 weeks, in order to understand the satisfaction of the case and the main caregiver on the interactive use of the App, a visual analog scale (visual analogy scale) composed of a parallel total length of 20 cm. analog scale), the score ranges from 0 to 100, with 0 representing overall dissatisfaction with the app's digital care plan, and 100 indicating overall satisfaction with the app's digital care plan. A line, and the corresponding score represents the satisfaction with the digital care plan after using the app for eight weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Hui Ping, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No